CLINICAL TRIAL: NCT03664479
Title: A Double-blind, Parallel Compensatory Medical Device Pivotal Clinical Study to Assess the Safety and Efficacy of the 4 Channel Neuromuscular Electrical Stimulation (NMES), Pilot Study
Brief Title: Assess the Safety and Efficacy of the 4 Channel NMES, Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: collected data showed significant difference in two groups.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-1706/402-001
Record Dates: First submitted 2018-04-06; First posted 2018-09-10 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-02

CONDITIONS: Dysphagia
Keywords: stroke; cervical spinal cord injury
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classical electrical stimulation protocol (Experimental): * apply 4 channel electrical stimulation device with protocol 1.
  * It will simultaneously stimulate suprahyoid, thyrohyoid and sternothyroid m with 4 channel electrical stimulation device.
  * during apply the device, we evaluate the manometry and videofluoroscopic swallowing study for evaluation of deglutition function.
  Interventions: Device: 4 channel Electrical Stimulation Device
- revised sequential activation protocol (Experimental): * apply 4 channel electrical stimulation device with protocol 2
  * Is a revised sequential activation protocol, it sequentially stimulate bilateral suprahyoid m (channel 1), pharyngeal constrictors (ch 2), thyrohyoid m (ch 3), sternothyroid m (ch 4) with 4 channel electrical stimulation device.
  * during apply the synchronized electrical stimulation device, we will evaluate the parameters same as group 1.
  Interventions: Device: 4 channel Electrical Stimulation Device

INTERVENTIONS:
Device: 4 channel Electrical Stimulation Device — electrical stimulation at muscles which related with deglutition

SUMMARY:
This study is a pilot study to prepare clinical trials to evaluate the safety and effectiveness of 4-channel electric stimulation therapy devices as a newly developed function for the treatment of dysphagia disorders.

The purpose of this study is to investigate the difference in effect by the electric stimulation method and to obtain the values such as mean, standard deviation and so on, and to determine the number of subjects to be studied for clinical trials of validation permission in the future.

DETAILED DESCRIPTION:
* Design: Prospective study
* Inclusion criteria of patient group: who has a dysphagia symptom and confirmed by video-fluoroscopic swallowing study(N=9)
* Intervention: Participants are divided into two group and applied electrical stimulation by a "Synchronized Electrical Stimulation Device(SESD)" in different protocol
* Main outcome measures: high-resolution manometry(HRM) parameters, videofluoroscopic parameters, EQ-5D (EuroQoL-5D) questionnaire

ELIGIBILITY:
Inclusion Criteria:

* patient who do not belong to the criteria excluded for subjects aged 19 years or older
* Patient who is confirmed to be dysphagia by videofluoroscopy
* Patients who need clinical application of electrical stimulation therapy equipment for dysphagia. ex) stroke, cervical spinal cord injury
* Those voluntarily agreeing to the clinical trial

Exclusion Criteria:

* Patient who refuse inspection, do not agree
* Simple "Commend obey", first step is impossible
* When instructions can not be executed due to dementia, psychiatric disorders, etc.
* Dysphagia occurs due to respiratory failure, neck surgery, etc.,
* Pregnant women and lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
pressure change | baseline/ change from baseline when electrical stimulation applied(the object of this study is to know the temporary change of dysphagia when stimulating with 4ch NMES.)
videofluoroscopic dysphagia scale | baseline/ change from baseline when electrical stimulation applied(the object of this study is to know the temporary change of dysphagia when stimulating with 4ch NMES.
  total score 100 from 0, 100 is worst outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jusuk Ryu, M.D. PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea